CLINICAL TRIAL: NCT01878201
Title: A Randomized, Double-blind, Valsartan 80 Mg-Referenced, Parallel Grouped, Therapeutic Exploratory Clinical Study to Evaluate the Antihypertensive Efficacy of Fimasartan 30 mg During 24 Hours in Patients With Mild to Moderate Essential Hypertension
Brief Title: A Valsartan 80 Mg-Referenced, Therapeutic Exploratory Clinical Study to Evaluate the Antihypertensive Efficacy of Fimasartan 30 mg During 24 Hours in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Seoul National University Bundang Hospital (Other); Kyungpook National University Hospital (Other); Chonnam National University Hospital (Other); Inje University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A657-BR-CT-L201
Record Dates: First submitted 2013-05-31; First posted 2013-06-14 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; 24 hours ABP monitoring(ABPM); antihypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fimasartan 30 mg (Experimental): Take one capsule filled with a Fimasartan 30 mg in the every morning
  Interventions: Drug: Fimasartan
- Valsartan 80 mg (Active Comparator): Take one capsule filled with a Valsartan 80 mg in the every morning
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Fimasartan — Fimasartan 30 mg
  Other Names: Kanarb
  Arms: Fimasartan 30 mg
Drug: Valsartan — Valsartan 80 mg
  Other Names: Diovan
  Arms: Valsartan 80 mg

SUMMARY:
The purpose of this study is to Evaluate the Antihypertensive efficacy of Fimasartan 30 mg during 24 hours in Patients with Mild to Moderate Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20 to 70 years
2. Essential hypertension subjects who are measured more 135/85 mmHg of average Diastolic Blood pressure (DBP) and Systolic Blood pressure (SBP) measured by ABP monitor at baseline visit(day 0)
3. Subjects who agreed to participate in this study and submitted the written informed consent
4. Subjects who considered to understand this study, be cooperative, and able to be followed-up whole of the study period

Exclusion Criteria:

1. Severe hypertension patients; more 180 mmHg of mean sitting SBP and/or more 110 mmHg of mean sitting DBP measured as an office Blood pressure (BP), before Randomization (Screening visit, Placebo run-in visit, Pre-Baseline visit, Baseline visit)
2. Patients with difference of office BP at selected one arm over DBP 10 mmHg and/or SBP 20 mmHg at screening visit
3. Patients with secondary hypertension
4. Patients with symptomatic orthostatic hypotension
5. Patients with severe insulin dependent or uncontrolled diabetes mellitus (HbA1c > 9%, increased regimen of oral hypoglycemic agent, using insulin at baseline visit)
6. Patients with severe heart disease, ischemic heart disease within 6 months, peripheral vascular disease, Percutaneous Transluminal Coronary Angiography (PTCA), Coronary Artery Bypass Graft (CABG)
7. Patients with significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia
8. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease
9. Patients with severe cerebrovascular disease within 6 months
10. Patients with known severe or malignancy retinopathy within 6 months
11. Patients with wasting disease, autoimmune disease, connective tissue disease
12. Patients with significant investigations - abnormal renal function (Creatinine more 1.5 times than upper limit of normal), abnormal liver function (Aspartate Transaminase(AST), Alanine Transaminase(ALT) more 2 times than upper normal)
13. Patients with surgical or medical disease which is able to be affect to absorption, distribution, metabolism, excretion
14. Patients with hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
15. Patients with significant investigations - Hypokalemia(Less than 3.5mmol/L), Hyperkalemia(exceeded 5.5mmol/L)
16. Patients with depletion of body fluid or sodium ion not able to correct
17. Patients with suspected or history of drug or alcohol abuse within the past two years
18. Childbearing, breast-feeding women and female who plan to become pregnancy or have a possibility of pregnancy but don't prevent conception with acknowledged methods
19. Patients with any chronic inflammation disease needed to chronic inflammation therapy
20. Patients with hepatitis type B or type C and carriers
21. Patients with laboratory test results indicating clinically significant abnormal results
22. Patients receiving medication that can affect blood pressure
23. Patients with history of allergic reaction to any angiotensin II antagonist
24. Patients with the medical histories of malignant tumor within 5years, except local basal cell carcinoma of the skin
25. Patients who took investigational drug within 12 weeks from screening visit or is going on the progress of other clinical trial
26. Subject who are judged unsuitable to participate in this study by investigator

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Mean Systolic Blood Pressure during 24 hours | 8 weeks from baseline visit
  To compare the difference of Mean Systolic Blood Pressure during 24 hours at 8 weeks from baseline visit

SECONDARY OUTCOMES:
Mean Diastolic Blood Pressure during 24 hours | 8 weeks from baseline visit
  To compare the difference of Mean Diastolic Blood Pressure during 24 hours at 8 weeks from baseline visit
Mean Diastolic Blood pressure and Systolic Blood pressure during daytime or nighttime | 8 weeks from baseline visit
  To compare the difference of Diastolic Blood pressure and Systolic Blood pressure during daytime or nighttime at 8 weeks from baseline visit
Sitting Diastolic Blood pressure and Systolic Blood pressure | 8 weeks from baseline visit
  To compare the difference of Sitting Diastolic Blood pressure and Systolic Blood pressure at 8 weeks from baseline visit
Trough-to-peak ratio | 8 weeks from baseline visit
  Trough-to-peak ratio of systolic blood pressure and diastolic blood pressure measured by ABP(Ambulatory Blood Pressure) monitor
Smoothness index | 8 weeks from baseline visit
  Smoothness index of systolic blood pressure and diastolic blood pressure measured by ABP monitor

OTHER OUTCOMES:
Adverse events | about 10~11weeks from placebo run-in visit
  Adverse evnt(AE)s are collected as a safety measure. All AEs are arranged based on severity, relevance to the investigational drug and serious adverse event each.
Adverse changes in laboratory test results | about 10~11weeks from screening visit
  Adverse changes in laboratory test results are collected as a safety measure. As a continuous data group for each test visit, adverse changes in laboratory test results present descriptive statistics (mean, standard deviation, minimum, maximum, etc.)
Adverse changes in electrocardiography(ECG) | about 10~11weeks from screening visit
  Adverse changes in ECG are collected as a safety measure. As a categorical data, adverse changes in ECG present frequency and percentage for each category.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-He Oh, professor, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea